CLINICAL TRIAL: NCT03210402
Title: REmodeling the Left Ventricle With Atrial Modulated Pacing
Acronym: REVAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REVAMP
Record Dates: First submitted 2017-02-27; First posted 2017-07-06 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Elevated night pacing on (Active Comparator)
  Interventions: Device: Elevated night pacing on
- Elevated night pacing off (Placebo Comparator)
  Interventions: Device: Elevated night pacing off

INTERVENTIONS:
Device: Elevated night pacing on — Device will be programmed to 100 beats per minute (bpm) for five hours during normal sleep times
  Arms: Elevated night pacing on
Device: Elevated night pacing off — Device will be programmed to normal lower rates
  Arms: Elevated night pacing off

SUMMARY:
New therapy tested in heart failure with preserved ejection fraction (HFpEF) patients with approved indications for pacing to determine if elevated pacing therapy is tolerated and whether there is a signal for efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had a market released dual chamber Medtronic Pacemaker with a Sleep function for at least 3 months
* Subject is stable on current medications
* Subject has dyspnea with exertion or diagnosed as New York Heart Association (NYHA) Class II or III Heart Failure
* Subject has had a prior Echo in past 6 months with: Ejection Fraction (EF) ≥ 50% and Diastolic volume <80 ml/m²
* Subject has evidence of hypertrophy (indexed to body surface area: men 115 g/m², women 95 g/m² or indexed to height: men 49.2 g/m2.7, women 46.7 g/m2.7) or Relative Wall thickness >0.42, or Wall Thickness>1.2cm (posterior wall)
* Subject is willing to sign and date the study Informed Consent Form (IC Form) - Subject is 18 years of age or older, or of legal age to give informed consent per local law
* Subject is expected to remain available for follow-up visits

Exclusion Criteria:

* Subject has permanent atrial fibrillation (AF) or AF noted on baseline interrogation rhythm strip
* Subject has uncontrolled BP; (systolic pressure needs to be >100 mmHg and <160 mmHg on medications)
* Subject has severe stenosis of the aortic or mitral valve, defined as valve area ≤1.0 cm² or severe regurgitation of the aortic or mitral valve
* Subject has symptomatic Chronic Obstructive Pulmonary Disease (COPD) requiring oxygen
* Subject's Pacemaker has less than 6 months of Pacemaker battery life
* Subject had an aortic valve replacement (surgical or TAVR) procedure less than 9 months prior to enrollment
* Subject's programmed upper rate limit is less than 100 bpm because of concerns of elevated pacing
* Subject is unable or unwilling to perform the 6 Minute Walk Test at all scheduled study visits
* Subject is currently enrolled or planning to enroll in a potentially confounding trial during the course of the study (co-enrollment in concurrent studies is only allowed when documented pre-approval is obtained from the Medtronic study manager)
* Subject is pregnant
* Subject meets any exclusion criteria required by local law
* Subject's life expectancy is less than 12 weeks
* Subject with medical condition that precludes the patient from participation in the opinion of the investigator
* Subject has known coronary disease with Class II angina

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Steinhaus, MD, Study Director — Medtronic CRHF
Locations (10):
- United States (10):
  - University of Arizona - Sarver Heart Center, Tucson, Arizona
  - St Joseph's Medical Center, Stockton, California
  - Northwestern University, Chicago, Illinois
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - The Lindner Research Center, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible subjects were approached for participation during the entire recruitment period (site activation through enrollment closure) at each participating site.
Pre-assignment Details: After completing a baseline visit but before randomization, all subjects received four weeks of elevated night pacing.
  8 subjects exited the study before randomization, and are not shown as exits in the study period table. Of these 8 subject exits, 3 exited after enrollment due to screening failures, and 5 exited between the baseline visit and randomization due to withdrawal by subject.
Groups:
- Pacing On: Elevated night pacing on: Device will be programmed to 100 beats per minute (bpm) for five hours during normal sleep times for 4 weeks, then therapy will be discontinued
- Pacing Off: Patient will receive no pacing therapy
Period: Overall Study
Arm/Group | Pacing On | Pacing Off
Started ((Randomization after baseline period)) | 9 | 5
Completed | 9 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Enrolled Patients: All enrolled patients
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex not collected for the 3 subjects who failed screening.
  Participants
    number analyzed (Participants) | 19
    Female | 8
    Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 22
NYHA Class [Count of Participants; unit: Participants] — NYHA = New York Heart Association
  Participants
    Classification not available | 4
    Subject Does Not have Heart Failure | 1
    Class 1)No symptoms and no limitation in ordinary physical activity | 0
    Class 2) Slight limitation of physical activity. | 9
    Class 3) Marked limitation of physical activity. | 8
    Class 4) Unable to carry on any physical activity without discomfort. Symptoms at rest. | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Remained on Study
Description: REVAMP is a Non-Significant Risk Investigation Device Exemption exploratory/feasibility study. The primary objective is to assess the feasibility of using the elevated night pacing intervention in subjects with heart failure with preserved ejection fraction. This primary objective does not involve statistical analysis, the number of participants that remained on study during each study phase were descriptively summarized.
Time Frame: Baseline through 12 week follow-up
Population: Subjects were randomized to these two arms after an initial 4-week baseline period in which all subjects had their device programmed to provide elevated night pacing.
Measure: Number; unit: participants
Arm/Group | Elevated Night Pacing on | Elevated Night Pacing Off
Number analyzed (Participants) | 9 | 5
participants | 9 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all patients from the time of enrollment through the time of study exit, which occurred 12 weeks after the baseline visit for subjects that did not exit early.
Description: Definitions are consistent with clinicaltrials.gov definitions.
Groups:
- Elevated Night Pacing On Before Randomization: This arm includes all subjects as assessed from study start until randomization at the 4-week visit. Note that all subjects received elevated night pacing during this period.
- Elevated Night Pacing On From Randomization To 8 Weeks: This arm includes subjects that were randomized to continue receiving elevated night pacing at the 4-week visit, as assessed from the 4-week visit to the 8-week visit.
- Elevated Night Pacing Off From Randomization To 8 Weeks: This arm includes subjects that were randomized to discontinue receiving elevated night pacing at the 4-week visit, as assessed from the 4-week visit to the 8-week visit.
- Elevated Night Pacing Off After 8 Weeks: This arm includes all subjects as assessed from the 8-week visit until study exit. Note that no subjects received elevated night pacing during this period.
Arm/Group | Elevated Night Pacing On Before Randomization | Elevated Night Pacing On From Randomization To 8 Weeks | Elevated Night Pacing Off From Randomization To 8 Weeks | Elevated Night Pacing Off After 8 Weeks
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/9 | 0/5 | 0/13
Serious Adverse Events (participants affected / at risk) | 4/22 | 1/9 | 2/5 | 0/13
Other Adverse Events (participants affected / at risk) | 9/22 | 1/9 | 0/5 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elevated Night Pacing On Before Randomization (N=22) | Elevated Night Pacing On From Randomization To 8 Weeks (N=9) | Elevated Night Pacing Off From Randomization To 8 Weeks (N=5) | Elevated Night Pacing Off After 8 Weeks (N=13)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elevated Night Pacing On Before Randomization (N=22) | Elevated Night Pacing On From Randomization To 8 Weeks (N=9) | Elevated Night Pacing Off From Randomization To 8 Weeks (N=5) | Elevated Night Pacing Off After 8 Weeks (N=13)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The patient after 25 mins of the pacemaker being programmed, she said "i don't feel well". she described slight chest pressure, she saw spots, and had a dizzy feeling.; Her blood pressure was unchanged
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study ended with fewer participants than was desired for the investigation. The study ended due to difficulty finding eligible patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participating Institution and Principal Investigator may publish the results of work performed under this Agreement, in accordance with the publication strategy described in the Protocol; provided, however, that any such Publication will be provided to Medtronic for review at least forty five (45) days prior to submission or presentation; provided, however, that such publication strategy in no way shall prevent Institution from freely utilizing data for Publication

DOCUMENTS (3):
  • Study Protocol (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03210402/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03210402/SAP_002.pdf
  • Informed Consent Form (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03210402/ICF_003.pdf